CLINICAL TRIAL: NCT07293598
Title: A Clinical, Histological, Cellular and Molecular Investigation of the Role of Fat and Inflammatory Cells in Melanoma Plasticity and Metastases
Brief Title: Investigation of the ROle of faT and inflAmmaTory Cells in mElanoma
Acronym: ROTATE
Status: Not yet recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp252
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Melanoma (Skin Cancer)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sample analysis only — Sample analysis only

SUMMARY:
This study is a retrospective, proof-of-concept sample study to investigate a novel histological finding within the primary melanoma tumour in a large population of melanoma patients to assess its prognostic significance.

This is a aims to validate the striking observation that a cross-talk between fat cells and leukocytes at the primary melanoma site promotes metastasis. In our unpublished pilot study, we have discovered an interesting finding whereby inflammatory cells extend from the tumour to and invading fat in the subcutaneous tissue and/or around the appendageal structures in the dermal skin in metastatic melanomas with distinct architectural changes within the fat. This finding was consistently present in metastatic and absent in non-metastatic melanomas. This new finding has both clinical and pathophysiological credence. Archival tissue blocks or human cell lines will be used in the first instance. As mitigation, experiments will be repeated with conditioned media obtained from co-culture of mixed primary immune cells obtained from peripheral blood mononuclear cell (PBMCs) and adipocytes induced from stem cells.

This study aims to:

* Investigate if the crosstalk between fat cells and tumour-infiltrating inflammatory cells defines the aggressiveness of primary cutaneous melanomas.
* Identify and perform biological spatial analysis of the inflammatory cells between the tumour and fat in the primary tumours.
* Investigate the interactions of fat cells and/or inflammatory cells in mediating melanoma cellular plasticity.

The patients have not provided consent and will be justified in this application

ELIGIBILITY:
Inclusion Criteria:

1. Melanomas treated between 1st January 2006 and 31st December 2015 OR
2. Patients treated at the Christie between 2014 and 2019.
3. Review of histological slides for presence or absence of relevant histological features.

   For group 3 and group 4:
4. Unique features of spitzoid melanomas

Exclusion Criteria:

* Inadequate slide quality
* Unable to view the entire cross section of the skin with the primary tumour hence, unable to assess the invasion of inflammatory cells into fat

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sample analysis of melanoma only
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
What is the predictive accuracy of inflammatory cell invasion into the subcutaneous fat layer in primary melanoma for determining the risk of metastasis and/or disease progression? | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided